CLINICAL TRIAL: NCT02193555
Title: Visual Performance of Prototype Contact Lens Designs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brien Holden Vision (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: CRTC2014-02
Record Dates: First submitted 2014-07-16; First posted 2014-07-17 (Estimated); Last update posted 2014-11-06 (Estimated); Status verified 2014-07

CONDITIONS: Presbyopia; Refractive Error
Keywords: Presbyopia; Refractive error correction; Contact lenses
MeSH Terms: conditions — Presbyopia; Refractive Errors

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non-presbyopic group (Other): Non-presbyopic group: age ranging from 7 to 39 years
  At each scheduled lens fitting visit, subjects will be allocated one pair of CLs to correct their refractive error. One pair of control (Acuvue 1- Day Moist, etafilcon A) or prototype (Iteration X, etafilcon A) CLs will be allocated for each lens fitting/assessment visit. Lenses will be worn for approximately 1 hour per visit.
  For each fitting visit, lenses will be fitted bilaterally.
  Interventions: Device: Etafilcon A, Senofilcon A
- Presbyopic group (Other): Presbyopic group: age 40 and above
  At each scheduled lens fitting visit, subjects will be allocated one pair of CLs to correct their refractive error. One pair of control (Acuvue Oasys for Presbyopia, senofilcon A) or prototype (Iteration X, etafilcon A) CLs will be allocated for each lens fitting/assessment visit. Lenses will be worn for approximately 1 hour per visit.
  For each fitting visit, lenses will be fitted bilaterally.
  Interventions: Device: Etafilcon A, Senofilcon A

INTERVENTIONS:
Device: Etafilcon A, Senofilcon A — 1 pair of either test or control lenses will be fitted on the subject for up to 1 hour of lens wear per visit (total of 2 fitting visits).
  Other Names: Control lenses; Non-presbyopic group; Brand name: 1-Day Acuvue® Moist®; Lens material: Etafilcon A; Presbyopic group; Brand name: Acuvue® Oasys® for Presbyopia; Lens material: Senofilcon A; Test lens; Brand name: Iteration X

SUMMARY:
The aim of this study is to assess the visual performance of prototype soft contact lens designs compared to a commercially available contact lens

DETAILED DESCRIPTION:
Prospective, participant-masked, randomised, stratified, crossover, bilateral wear, dispensing clinical trial where participants will wear the prototype (test) and the commercial (control) lens. A minimum of an overnight washout period is required between the fitting /assessment visits.

ELIGIBILITY:
Inclusion Criteria:

* Able to read and comprehend English and give informed consent as demonstrated by signing a record of informed consent.
* Be at least 7 years old, male or female.
* Willing to comply with the wearing and clinical trial visit schedule as directed by the Investigator.
* Have ocular health findings considered to be "normal" and which would not prevent the participant from safely wearing contact lenses.
* Correctable to at least 6/12 (20/40) or better with both eyes with contact lenses.
* Be suitable and willing to wear contact lenses.

Exclusion Criteria:

* Any pre-existing ocular irritation, injury or condition (including infection or disease) of the cornea, conjunctiva or eyelids that would preclude contact lens fitting and safe wearing of contact lenses.
* Any systemic disease that adversely affects ocular health e.g. diabetes, Graves' disease, and auto immune diseases such as ankylosing spondylitis, multiple sclerosis, Sjögrens syndrome and systemic lupus erythematosus. Conditions such as systemic hypertension and arthritis do not automatically exclude prospective participants.
* Use of or a need for concurrent category S3 and above ocular medication at enrolment and/or during the clinical trial.
* Use of or a need for any systemic medication or topical medications which may alter normal ocular findings / are known to affect a participant's ocular health / physiology or contact lens performance either in an adverse or beneficial manner at enrolment and/or during the clinical trial.
* Eye surgery within 12 weeks immediately prior to enrolment for this trial.

NB: Systemic antihistamines are allowed on an "as needed basis", provided they are not used prophylactically during the trial and at least 24 hours before the clinical trial product is used.

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2014-07; Primary Completion 2014-09 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Visual performance | After about 20 minutes of lens wear
  Visual acuity

SECONDARY OUTCOMES:
Subjective responses | After about 40 minutes of lens wear
  Subjective ratings of vision

CONTACTS AND LOCATIONS:
Overall Officials: Jiyoon Chung, BOptom, Principal Investigator — Brien Holden Vision Institute
Locations (1):
- Brien Holden Vision Institute, Clinical Research Trials Center, Sydney, New South Wales, Australia

REFERENCES:
- [Background] Morgan PB, Efron N. A decade of contact lens prescribing trends in the United Kingdom (1996-2005). Cont Lens Anterior Eye. 2006 May;29(2):59-68. doi: 10.1016/j.clae.2006.02.008. Epub 2006 Mar 31. PMID 16580247
- [Background] Stapleton F, Keay L, Edwards K, Naduvilath T, Dart JK, Brian G, Holden BA. The incidence of contact lens-related microbial keratitis in Australia. Ophthalmology. 2008 Oct;115(10):1655-62. doi: 10.1016/j.ophtha.2008.04.002. Epub 2008 Jun 5. PMID 18538404
- [Background] Anstice NS, Phillips JR. Effect of dual-focus soft contact lens wear on axial myopia progression in children. Ophthalmology. 2011 Jun;118(6):1152-61. doi: 10.1016/j.ophtha.2010.10.035. Epub 2011 Jan 26. PMID 21276616
- [Background] Sankaridurg P, Holden B, Smith E 3rd, Naduvilath T, Chen X, de la Jara PL, Martinez A, Kwan J, Ho A, Frick K, Ge J. Decrease in rate of myopia progression with a contact lens designed to reduce relative peripheral hyperopia: one-year results. Invest Ophthalmol Vis Sci. 2011 Dec 9;52(13):9362-7. doi: 10.1167/iovs.11-7260. PMID 22039230